CLINICAL TRIAL: NCT06875635
Title: Effect of Pelvic Floor Muscle Training on Pelvic Floor Dysfunction and Quality of Life in Patient Undergoing Gynecological Surgery
Brief Title: Pelvic Floor Dysfunction and Quality of Life in Patient Undergoing Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Majida zaffar
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Floor Dysfunction
Keywords: pelvic floor training ,; gynecological surgery,; quality of life,; strength of pelvic floor muscle
MeSH Terms: interventions — Lead

STUDY DESIGN:
Intervention Model Description: There will be comparison between 3 groups.Two intervention group and 1 control group
Who Masked: Investigator
Masking Description: The Principal investigator or the researcher will be kept blind about the group allocation and intervention or assessment of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prepost PFMT Group (Experimental): Routine medical care and pre & post-op - op protocol of pelvic floor muscle training .1 month prior and 8 weeks post op protocol in patient undergoing gynecological surgery
  Interventions: Other: Pre and Post op pelvic floor muscle training
- Post PFMT Group (Experimental): Only Post-op pelvic floor muscle training for 8 weeks along with Routine medical care
  Interventions: Other: Only post op pelvic floor muscle training
- Control (Other): Routine medical care was given
  Interventions: Other: Routine medical care

INTERVENTIONS:
Other: Pre and Post op pelvic floor muscle training — pre op exercises: Breathing exercise ,Kegel exercise ,Abdominals exercise include pelvic tilt ,knee rolling with abdominal contraction post op exercise :breathing exercise, circulatory exercise i.e ankle pump and heel slides, and bed mobility along with pre op exercise
  Arms: Prepost PFMT Group
Other: Only post op pelvic floor muscle training — post op exercise :breathing exercise, circulatory exercise i.e ankle pump and heel slides, and bed mobility along with pre op protocol
  Arms: Post PFMT Group
Other: Routine medical care — Circulatory exercise Breathing exercise Administrating analgesic Nursing care
  Arms: Control

SUMMARY:
The purpose of the study is to assess the pelvic floor dysfunction and quality of life in patient undergoing gynecological surgery.Common gynecological surgeries done for prolapse, fibroids, and cervical abnormality and also for Gynecological cancer.Early physiotherapy after gynecological surgery improves recovery by managing pain, restoring movement, and strengthening muscles, especially the pelvic floor.Conservative treatments like pelvic floor muscle exercises, biofeedback, and lifestyle changes can help with pelvic symptoms, including urinary incontinence and mild to moderate prolapse.

DETAILED DESCRIPTION:
This is a randomized control trial to see the effects of pelvic floor training on pelvic floor dysfunction and quality of life in patient undergoing gynecological surgery. Females meeting the inclusion and exclusion criteria will be divided into three groups by convenient sampling technique. A sample size of 48 females with 16 females in each group. Group A will be treated four weeks pre and 8 weeks post op pelvic floor training exercises, group B will be treated only 8 weeks post op pelvic floor training exercises and group C will receive basic post op nursing care. Group A and B will have three treatment sessions per week Assessment will be done at 0 week (1month prior to surgery), 1 day before surgery, 2nd , 4th, 6th and 8th week after surgery. Females will be screened by Pelvic organ distress inventory (PFDI-20) and Pelvic floor impact questionnaire (PFIQ-7).

ELIGIBILITY:
Inclusion Criteria:

* Women age:40 -60yrs
* undergoing vaginal or laparoscopic-assisted vaginal surgery for either POP repair (primary or recurrent), and/or hysterectomy

Exclusion Criteria:

* Emergency Surgery
* Chronic Illness
* Unstable Mental State

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only female
Enrollment: 48 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Pelvic organ distress inventory (PFDI-20) | From Baseline to 1 day prior to surgery, 2nd,4th,6th and 8th week of intervention
  Pelvic floor Distress inventory questionnaire is comprised of 3 Sections, including pelvic organ prolapse distress inventory (POPDI-6) from question 1 to 6, urinary distress inventory (UDI-6) from questions 7-12 and colorectal anal distress inventory (CRADI-8) from questions 13-20.
  The total score ranges from 0 to 300, with higher scores indicating greater distress.the ICC value of the tool is 0.93
Pelvic floor impact questionnaire (PFIQ-7) | From Baseline to 1 day prior to surgery, 2nd,4th,6th and 8th week of intervention
  The pelvic floor impact questionnaire is used for quality of life assessment. it has 3 sections, including Urinary impact questions, Colorectal anal impact questions, and Pelvic organ prolapse impact questionnaire. The total score ranges from 0-300. The ICC value of PFIQ is 0.77

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PhD, Principal Investigator — Riphah International University, Islamabad, Pakistan
Locations (1):
- Lady Reading Hospital MTI, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No